CLINICAL TRIAL: NCT03105596
Title: Study of Chidamide Plus DICE Regimen for Patients With Relapse or Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Chidamide Plus DICE Regimen for Patients With Relapse or Refractory B-cell Non-Hodgkin's Lymphoma (NHL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chidamide plus DICE
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide plus DICE regimen (Experimental): Chidamide combined with DICE (Dexamethasone, Ifosfamide, Cisplatin and Etoposide) regimen
  Interventions: Drug: Chidamide plus DICE Regimen

INTERVENTIONS:
Drug: Chidamide plus DICE Regimen — Chidamide 20mg orally d1, 4, 8, 11, 15, 18; Dexamethasone 10mg，ivg, d1-4; ifosfamide 1g/m2, ivg, d1-4, given over 4 hours; Mesna 0.4g, 0,4,8,12 hours during Ifosfamide transfusion, ivg, d1-4; Cisplatin 25mg/m2, ivg, d1-4; Etoposide 60mg/m2, ivg. d1-4.

SUMMARY:
This is a prospective phase II clinical trial to observe the efficacy and safety of Chidamide combined with DICE (Dexamethasone, Ifosfamide, Cisplatin and Etoposide) in patients with relapsed or refractory B-cell Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
Chidamide，a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. The aim of this study was to observe the efficacy and safety of Chidamide combined with DICE in patients with relapsed or refractory B-cell Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as B-cell Non-Hodgkin's Lymphoma (NHL) according to "2008 WHO classification of tumors of haematopoietic and lymphoid tissues", including Diffuse Large B-Cell Lymphoma, Follicular Lymphoma, Mantle Cell Lymphoma, Marginal Zone Lymphoma, transformed indolent lymphoma, and other subtypes that investigators consider to be appropriate to be enrolled;
2. Patients must have received at least one systemic treatment (including chemotherapy), but did not achieve remission or had relapse after remission;
3. At least one measurable lesion;
4. Age18-65 years, male or female; ECOG performance status 0-1;
5. Without bone marrow involvement. Blood routine test: absolute neutrophil count ≥1.5 × 109/L, platelet ≥100 × 109/L, Hb ≥ 90g/L;.
6. Life expectancy no less than 3 months;
7. Not received chemotherapy, targeted medicine or stem cell transplantation 4 weeks before enrollment;
8. Patients have signed the Informed Consent Form.

   -

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures.
2. QTc elongation with clinical significance ( male˃ 450ms, female˃ 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment;
3. pericardial effusion ≥10mm sum of echo-free spaces by echocardiography;
4. Patients have undergone organ transplantation;
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment.
6. Patients with active hemorrhage.
7. Patients with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction.
8. Patients with active infection, or with continuous fever within 14 days prior to enrollment.
9. Patients with active infection of HBV, HCV or HIV;
10. Had major organ surgery within 6 weeks prior to enrollment.
11. Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum).
12. Patients with mental disorders or those do not have the ability to consent.
13. Patients with drug abuse, long term alcoholism that may impact the results of the trial.
14. Patients who have central nervous system involvements;
15. Non-appropriate patients for the trial according to the judgment of the investigators.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-04-11 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | every 6 weeks until 2 years
  the total proportion of patients with complete response（CR or CRu）and partial response（PR）

SECONDARY OUTCOMES:
progression-free survival（PFS） | 2 years
  Time from treatment until disease progression or death
events-free survival（EFS） | 2 years
  Time from treatment to disease progression, death, or discontinuation of treatment for any reason
overall survival（OS） | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Undecided